CLINICAL TRIAL: NCT07191613
Title: Effects of the HAPPY GO GO Somatosensory Game on Physical and Mental Health of Rural Community-Dwelling Elderly
Brief Title: Effects of HAPPY GO GO Game on Health of Rural Elderly
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chang Gung University of Science and Technology (Other)
Collaborators: National Science and Technology Council, Taiwan (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 114-0548
Record Dates: First submitted 2025-08-29; First posted 2025-09-25 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2025-09

CONDITIONS: Frailty at Older Adults; Health Promotion
Keywords: Somatosensory Game; Community-Dwelling Elderly; Mental Health
MeSH Terms: conditions — Psychological Well-Being

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HAPPY GO GO Exergame (Experimental): Participants in the intervention group will engage in the "HAPPY GO GO" somatosensory exergame program. The intervention consists of structured game-based physical activity sessions, conducted once per week for a total duration of 12 weeks. Each session includes interactive, movement-based tasks designed to promote physical health, and mental well-being among community-dwelling older adults.
  Interventions: Behavioral: HAPPY GO GO Somatosensory Game
- Usual Daily Activities (No Intervention): Participants in the control group will not receive the game-based intervention. They will continue with their usual daily activities without structured exercise sessions. Health outcomes will be assessed at baseline and post-intervention for comparison with the experimental group.

INTERVENTIONS:
Behavioral: HAPPY GO GO Somatosensory Game — Participants in the intervention group will engage in the "HAPPY GO GO" somatosensory exergame program. The intervention consists of structured game-based physical activity sessions, conducted once per week for a total duration of 12 weeks. Each session includes interactive, movement-based tasks designed to promote physical health, and mental well-being among community-dwelling older adults.
  Arms: HAPPY GO GO Exergame

SUMMARY:
The goal of this quasi-experimental clinical trial is to evaluate the effects of the "HAPPY GO GO" somatosensory game on physical and mental health in community-dwelling older adults aged 65 years and above living in rural Chiayi County, Taiwan. The main questions it aims to answer are:

* Does participation in the somatosensory game improve physical health outcomes (e.g., balance, mobility, functional fitness)?
* Does participation improve mental health outcomes (e.g., mood, depressive symptoms)? Researchers will compare an intervention group, which participates in the game-based exercise program, with a control group that does not receive the intervention, to evaluate changes in health status.

Participants in the intervention group will take part in structured game-based physical activity sessions over several weeks, designed to promote engagement, improve physical performance, and support psychological well-being.

ELIGIBILITY:
Inclusion Criteria:

* Community-dwelling older adults aged 65 years or above living in rural areas of Chiayi County, Taiwan.
* Clear consciousness and able to communicate in Mandarin or Taiwanese.
* Willing to provide informed consent and participate in the study procedures.

Exclusion Criteria:

* Not actually residing in the community.
* Unable to comply with the intervention program.
* Cognitive impairment or inability to cooperate with data collection.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2025-08-21 (Actual); Primary Completion 2026-01-31 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Change in Frailty Status | Baseline and 12 weeks after intervention
  Frailty will be assessed using the Study of Osteoporotic Fractures (SOF) Index, which consists of three items commonly used in Taiwan's Ministry of Health and Welfare community frailty screening program. The SOF Index has a score range from 0 to 3, where a higher score indicates greater frailty (worse outcome).
  Score = 0: Robust Score = 1: Pre-frail Score = 2-3: Frail
Change in Lower Limb Flexibility | Baseline and 12 weeks after intervention
  Flexibility of the lower limbs will be assessed using the chair sit-and-reach test. Higher scores (in centimeters) indicate better flexibility.
Change in Upper Limb Flexibility | Baseline and 12 weeks after intervention.
  Flexibility of the upper limbs will be assessed using the back scratch test. Higher scores (in centimeters) indicate better flexibility.
Change in Agility and Dynamic Balance | Baseline and 12 weeks after intervention
  Agility and dynamic balance will be assessed using the 2.44-meter timed up-and-go test. Shorter times indicate better performance.
Change in Muscle Strength | Baseline and 12 weeks after intervention
  Muscle strength will be assessed using the 30-second chair stand test (lower limb strength) and the 30-second biceps curl test (upper limb strength, 8 lbs men / 5 lbs women). Higher repetitions indicate better strength.
Change in Cardiopulmonary Endurance | Baseline and 12 weeks after intervention
  Cardiopulmonary endurance will be measured using the 2-minute step test. Higher step counts indicate better endurance.

OTHER OUTCOMES:
Change in Body Mass Index (BMI) | Baseline and 12 weeks after intervention
  BMI will be calculated from measured height and weight using a standardized anthropometric assessment.

CONTACTS AND LOCATIONS:
Locations (1):
- Chang Gung University of Science and Technology, Chiayi Campus, Chiayi City, Taiwan

IPD SHARING:
Plan to Share IPD: No